CLINICAL TRIAL: NCT01218932
Title: Phase 1, Open-Label Study to Evaluate Potential Pharmacokinetic Interaction of Orally Administered Primaquine and Chloroquine in Healthy Thai Adult Subjects
Brief Title: Pharmacokinetic Study of Primaquine and Chloroquine in Healthy Subjects
Acronym: PQCQ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FTM1001
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Vivax Malaria
Keywords: primaquine; chloroquine; pharmacokinetic; interactions
MeSH Terms: conditions — Malaria, Vivax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Primaquine only, followed by chloroquine/primaquine, followed by chloroquine only
  Interventions: Drug: A
- B (Active Comparator): Primaquine alone, followed by chloroquine, followed by chloroquine/primaquine
  Interventions: Drug: B

INTERVENTIONS:
Drug: A — Subjects in A group who receive regimen 1 of primaquine (PQ) on the first admission (visit 2) will receive regimen 2 of primaquine and chloroquine combination (PQ and CQ) on second admission (visit 3) after 1 week wash out period and will finish with regimen 3 of Chloroquine (CQ) on the third admission (visit 4) after 8 weeks wash out period.
  Arms: A
Drug: B — Subjects in B group who receive regimen 1 of primaquine ( PQ) will receive regimen 2 of chloroquine (CQ) on second admission (visit 3) after 1 week wash out period and regimen 3 of primaquine and chloroquine combination (PQ and CQ)on third admission( visit 4) with 8 week wash out period in between.
  Arms: B

SUMMARY:
This is a standard pharmacokinetic interaction study. Subjects will be randomized to be either group A or B. Group A. Subjects will have 3 hospitalizations to complete. Each hospitalization will be about 12-24 hours depends on each regimen. Subjects in A group who receive regimen 1 of primaquine (PQ) on the first admission (visit 2) will receive regimen 2 of primaquine and chloroquine combination (PQ and CQ) on second admission (visit 3) after 1 week wash out period and will finish with regimen 3 of Chloroquine (CQ) on the third admission (visit 4) after 8 weeks wash out period.

Subjects in B group who receive regimen 1 of primaquine (PQ) will receive regimen 2 of chloroquine (CQ) on second admission (visit 3) after 1 week wash out period and regimen 3 of primaquine and chloroquine combination (PQ and CQ)on third admission(visit 4) with 8 week wash out period in between.

DETAILED DESCRIPTION:
Chloroquine and primaquine, has been first therapy for Plasmodium vivax and ovale malaria for over 50 years, and has been part of National policy in Thailand for decades. Primaquine is the only available hypnozoitocidal drug for P.vivax and gametocytocidal agent for Plasmodium falciparum malaria. Despite this enormous use knowledge about the mechanism of activity, pharmacokinetic properties, resistance and toxicity of primaquine are limited. Primaquine at the previously used dose for radical cure (15 mg base/day for 14 days) is also weakly effective against asexual stages of P. vivax malaria [4] The higher dose of 30 mg daily evaluated for malaria prophylaxis is now also generally recommended for radical cure. In the standard radical cure regimen, primaquine is usually given after the 3-day course of chloroquine, but there has been no study to inform timing of dosing so this decision is arbitrary. Despite the multistage specificity against the malaria parasite, and extensive recommendations, primaquine is currently underused because of uncertainties over safety, efficacy and dosage. Primaquine is an oxidant drug and causes haemolysis in patients with glucose-6-phosphate dehydrogenase deficiency (G6PD). Although several studies of the metabolites of the primaquine and chloroquine have been conducted over the past few years remarkably little is known about the interaction between these two commonly coadministered drugs.

This study is open-label pharmacokinetic study. Healthy 16 volunteers will be recruited to the established volunteer facility at single site at the Hospital for Tropical Diseases to determine the pharmacokinetic properties of primaquine and it's main active metabolites and evaluate any interaction with chloroquine.in order to provide clinical guidance for the optimum primaquine/chloroquine treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as judged by a responsible physician with no abnormality identified on a medical evaluation including medical history and physical examination.
2. Males and Females aged between 18 years to 60 years.
3. A female is eligible to enter and participate in this study if she is: of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy or of childbearing potential, has a negative serum pregnancy test at screening and urine pregnancy test prior to start the study drug in each period, and abstain from sexual intercourse or agrees to using effective contraceptive methods (e.g., intrauterine device, hormonal contraceptive drug, tubal ligation or female barrier method with spermicide) during the study until completion of the follow-up procedures
4. A male is eligible to enter and participate in this study if he: agrees to abstain from (or use a condom during) sexual intercourse with females of childbearing potential or lactating females; or is willing to use a condom/spermicide, during the study until completion of the follow-up procedures.
5. Read, comprehend, and write at a sufficient level to complete study-related materials.
6. Provide a signed and dated written informed consent prior to study participation.
7. Normal electrocardiogram (ECG) with QTc <450 msec.
8. Willingness and ability to comply with the study protocol for the duration of the trial.

Exclusion Criteria:

1. Females who are pregnant, trying to get pregnant, or are lactating.
2. The subject has evidence of active substance abuse that may compromise safety, pharmacokinetics, or ability to adhere with protocol instructions.
3. A positive pre-study hepatitis B surface antigen, positive hepatitis C antibody, or positive human immunodeficiency virus-1 (HIV-1) antibody result at screening.
4. Subjects with a personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de points (heart failure, hypokalemia).
5. Subjects with a family history of sudden cardiac death.
6. A creatinine clearance <70 mL/min as determined by Cockcroft-Gault equation:

   CLcr (mL/min) = (140 - age) * Wt / (72 * Scr) (multiply answer by 0.85 for females) Where age is in years, weight (wt) is in kg, and serum creatinine (Scr) is in units of mg/dL [Cockcroft, 1976].
7. History of alcohol or substance abuse or dependence within 6 months of the study: History of regular alcohol consumption averaging >7 drinks/wk for women or >14 drinks/wk for men. One drink is equivalent to 12 g alcohol = 5 oz (150 mL) of wine or 12 oz (360 mL) of beer or 1.5 oz (45 mL) of 80 proof distilled spirits within 6 months of screening.
8. Use of prescription or non-prescription drugs except paracetamol at doses of up to 2 grams/day, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until the completion of the follow-up procedure, unless in the opinion of investigator, the medication will not interfere with the study procedures or compromise subject safety; the investigator will take advice from the manufacturer representative as necessary.
9. The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication.
10. The subject is unwilling to abstain from ingesting alcohol within 48 hours prior to the first dose of study medication until collection of the final pharmacokinetic sample during each regimen.
11. Subjects who have donated blood to the extent that participation in the study would result in more than 300 mL blood donated within a 30-day period. Note: This does not include plasma donation.
12. Subjects who have a history of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the trial. In addition, if heparin is used during pharmacokinetic sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
13. Subjects with unstable medical conditions that, in the opinion of the investigator would compromise their participation in the trial
14. Those who, in the opinion of the investigator, have a risk of non-compliance with study procedures.
15. Lack of suitability for participation in this study, for any reason, in the opinion of the investigator.
16. AST or ALT >1.5 upper limit of normal (ULN)
17. Subjects with history of renal disease, hepatic disease, and/or cholecystectomy
18. G6PD deficient.
19. Abnormal methaemoglobin level.
20. Subjects who have anemia, Hb <12 for both male and female
21. History of malaria treatment with Primaquine and/or Chloroquine within 12 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
AUC | 36 days
  Area under the plasma concentration time AUC 0-∞curve for primaquine and metabolites (mPQ) when given alone and together with chloroquine

SECONDARY OUTCOMES:
Cmax | 36 days
  Primaquine and metabolites maximum concentrations, chloroquine and metabolites maximum concentration and AUC
Elimination rate | 36 days
  Primaquine and metabolites (mPQ) elimination rate constants (mPQ-λz), and elimination half life (mPQ-t1/2),chloroquine metabolite(s) elimination rate constant (mCQ-λz), and elimination half life (mCQ-t1/2)
Adverse events | 36 days
  Safety and tolerability parameters, including adverse events, clinical laboratory, and vital signs assessments
Pharmacogenetics | 36 days
  Pharmacogenetic polymorphisms in the case of unusually high or low drug levels

CONTACTS AND LOCATIONS:
Overall Officials: Podjanee Jittamala, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Hospital For Tropical Diseases, Bangkok, Thailand

REFERENCES:
- [Derived] Pukrittayakamee S, Tarning J, Jittamala P, Charunwatthana P, Lawpoolsri S, Lee SJ, Hanpithakpong W, Hanboonkunupakarn B, Day NP, Ashley EA, White NJ. Pharmacokinetic interactions between primaquine and chloroquine. Antimicrob Agents Chemother. 2014 Jun;58(6):3354-9. doi: 10.1128/AAC.02794-13. Epub 2014 Mar 31. PMID 24687509